CLINICAL TRIAL: NCT06087276
Title: Phase 3, Decentralized, Randomized, Double-Blind, Placebo Controlled, Parallel Design, Randomized Withdrawal, and Long-term Safety Study to Evaluate the Efficacy and Safety of Ulixacaltamide (PRAX-944) in Adults With Essential Tremor
Brief Title: Essential 3 - Decentralized, Phase 3 Study Evaluating the Safety and Efficacy of Ulixacaltamide in Essential Tremor (ET)
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRAX-944-321
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Essential Tremor
Keywords: Movement Disorder; Benign Essential Tremor; Familial Tremor; Hereditary Essential Tremor; Movement Disorder Agents; Calcium Channels, T-type
MeSH Terms: conditions — Essential Tremor; Movement Disorders

STUDY DESIGN:
Intervention Model Description: * Parallel Design: A 12-week parallel design (PD) randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of ulixacaltamide compared with placebo.
  * Randomized Withdrawal: A 12-week randomized withdrawal (RW), double-blind, placebo-controlled study to evaluate the efficacy, maintenance of response, and durability of effect in participants who respond to ulixacaltamide and safety.
  * Long-term Safety Study: A LTSS study to evaluate the long-term safety of ulixacaltamide for up to approximately 3 years. The first 2 weeks of the LTSS will be double-blind.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded randomization into either the Parallel Design or Randomized Withdrawal studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Parallel Design: ulixacaltamide arm (Experimental): Double-blind Part: Oral dosing, once daily in the morning with titration over 14 days to 60 mg ulixacaltamide: 7 days of 20 mg, 7 days of 40 mg, 70 days of 60 mg
  Interventions: Drug: 60 mg ulixacaltamide
- Parallel Design: placebo arm (Placebo Comparator): Double-blind Part: Oral dosing, once daily in the morning: 84 days of placebo
  Interventions: Drug: Placebo
- Randomized Withdrawal (Experimental): Double-blind Part: Oral dosing, once daily in the morning with titration over 14 days to 60 mg ulixacaltamide: 7 days of 20 mg, 7 days of 40 mg, 42 days of 60 mg
  Randomized Withdrawal Part: Following double-blind part: 1:1 randomization to placebo or 60 mg ulixacaltamide for 28 days
  Interventions: Drug: 60 mg ulixacaltamide; Drug: Placebo
- Long-term Safety Study: Essential1 rollovers (Experimental): Open-label Part: Oral dosing, once daily in the morning up to 3 years 60 mg ulixacaltamide
  Interventions: Drug: 60 mg ulixacaltamide
- Long-term Safety Study: Parallel Design and Randomized Withdrawal rollovers (Experimental): Open-label Part for patients previously on placebo: Oral dosing, once daily in the morning with titration over 14 days to 60 mg ulixacaltamide: 7 days of 20 mg, 7 days of 40 mg, up to 3 years 60 mg ulixacaltamide
  Open-label Part for patients previously on 60 mg ulixacaltamide: Oral dosing, once daily in the morning up to 3 years 60 mg ulixacaltamide
  Interventions: Drug: 60 mg ulixacaltamide
- Long-term Safety Study: Direct Enrollment to LTSS Study (Experimental): Oral dosing, once daily in the morning with titration over 14 days to 60 mg ulixacaltamide: 7 days of 20 mg, 7 days of 40 mg, up to 3 years 60 mg ulixacaltamide
  Interventions: Drug: 60 mg ulixacaltamide

INTERVENTIONS:
Drug: 60 mg ulixacaltamide — Once daily oral treatment with titration
  Arms: Long-term Safety Study: Direct Enrollment to LTSS Study; Long-term Safety Study: Essential1 rollovers; Long-term Safety Study: Parallel Design and Randomized Withdrawal rollovers; Parallel Design: ulixacaltamide arm; Randomized Withdrawal
Drug: Placebo — Once daily oral treatment
  Arms: Parallel Design: placebo arm; Randomized Withdrawal

SUMMARY:
The goal of this clinical study is to compare ulixacaltamide and placebo treatment in essential tremor. The main question it aims to answer is:

• Is ulixacaltamide a safe and efficacious treatment for patients with essential tremor?

Participants will be asked to participate in one of two clinical studies where they will be treated with either ulixacaltamide or placebo for a period of up to 12 weeks. After the controlled study completion, they will be eligible to participate in a long-term, open-label safety study (LTSS) and be treated with ulixacaltamide. Participants are eligible to enroll directly into the LTSS if they previously participated in an essential tremor trial, received sponsor invitation after being deemed ineligible for the controlled study, or following enrollment closure of the controlled study.

DETAILED DESCRIPTION:
PRAX-944-321 is a decentralized, Phase 3, multi-study, clinical trial evaluating the safety and efficacy of ulixacaltamide in essential tremor (ET). The study includes 3 separate and simultaneous phase 3 pivotal studies where all participants undergo one screening process. The first study is a parallel design (PD) enrolling approximately 400 patients, the second is a randomized withdrawal (RW) enrolling approximately 200 patients and the last is a long-term safety study (LTSS) comprising up to 1000 patients.

A total of 4 key efficacy hypotheses are being tested prospectively in the study. The analysis will be conducted simultaneously, with unblinding only occurring once. Hypotheses - 1) how do patients compare between ulixacaltamide and placebo after 56 days of intervention in the PD study, 2) for patients exposed to ulixacaltamide in the RW study who improved by at least 3 points in the mADL11 scale, which proportion maintains response after randomization staying on ulixacaltamide compared to placebo after re-randomization at day 56, 3) how does the pooled group of patients receiving ulixacaltamide in both studies (PD and RW) compare to placebo patients from the parallel design study after 56 days of intervention, 4) how do patients receiving ulixacaltamide in the RW study compare to placebo patients from the PD study after 56 days of intervention.

ELIGIBILITY:
Inclusion Criteria for Study 1 PD and Study 2 RW:

1. Has a body mass index (BMI) at Screening of ≥18 kg/m2.
2. Has a clinical diagnosis of ET confirmed during screening and characterized by postural and action tremor.
3. If currently receiving medication prescribed for ET, must be on ≤1 medications, on stable dose(s) for at least 1 month prior to Screening, and willing to maintain stable dose(s) throughout the study. As needed (PRN) use of prescribed ET medicines is not allowed with the exception of propranolol PRN. Participants prescribed propranolol PRN are eligible but must discontinue the PRN dose after the first day of screening. Primidone use is not allowed within 2 weeks prior to screening and throughout duration of study.
4. Women of childbearing potential must undertake pregnancy tests, with a documented negative serum pregnancy test at Screening, negative urine pregnancy tests at Baseline (Day 1) prior to administration of study drug, throughout the intervention periods (as outlined in the SoA) and at the SFU or ED Visit, as appropriate.
5. Is willing and able to use contraception as defined in the protocol and ICF.
6. Has been assessed as an appropriate and suitable candidate by investigator and has a neurological exam and medical record(s) consistent with ET diagnosis, as confirmed by the ERC central reviewer.
7. Confirm key inclusion criteria at Baseline

Exclusion Criteria for Study 1 PD and Study 2 RW:

1. Neuropathy, muscle weakness, arthropathy or other musculoskeletal diagnosis of the upper extremity that impairs dexterity or function.
2. Has a known hypersensitivity to any component of the formulation of ulixacaltamide.
3. Is unwilling or unable to refrain from episodic use of medication(s)/substance(s) that might interfere with the evaluation of tremor during the study.
4. Is sporadically using a benzodiazepine, sleep medication or anxiolytic (as further defined in the protocol), that in the judgement of the investigator or sponsor would confound the assessment of tremor.
5. Has trauma to the nervous system within 3 months preceding the onset of tremor.
6. Has a history of unilateral tremor or clinical evidence of another medical, neurological, or psychiatric condition that may explain or cause tremor, including but not limited to Parkinson's disease, Huntington's disease, Alzheimer's disease, stroke with neurologic sequelae, intention tremor (IT) caused by etiology other than ET, cerebellar disease (including spinocerebellar ataxias), primary dystonia, Fragile X Tremor/Ataxia syndrome or family history of Fragile X syndrome, traumatic brain injury, psychogenic tremor, alcohol or benzodiazepine abuse or withdrawal, multiple sclerosis, polyneuropathy (diabetic neuropathy allowed if disease does not affect gait or balance and does not involve upper extremity), and endocrine states such as uncontrolled or inadequately treated hypothyroidism, food, or supplement induced movement disorders (e.g., tremor related to beta agonists or caffeine), or other medical, neurological, or psychiatric conditions that may explain or cause tremor.
7. Has had prior magnetic resonance-guided focused ultrasound or surgical intervention for ET such as a deep brain stimulator (DBS) or lesion therapy such as thalamotomy.
8. Has had botulinum toxin injection for ET in the 6 months prior to Screening or throughout the study.
9. Is using the Cala trio health device for ET in 14 days prior to Screening or throughout the study.
10. Is unwilling or unable to refrain from drinking alcohol 24 hours before and during clinical study assessments, or regular use of alcohol that would preclude abstinence from alcohol for this time period around visits.
11. Has a history of substance use disorder consistent with Diagnostic and Statistical Manual of Mental Disorders Fifth Edition Text Revision (DSM-5-TR) criteria. Participants with a previous diagnosis of substance use disorder who have been in remission for at least 2 years can participate in the study.
12. Is currently pregnant or breastfeeding or is planning to become pregnant during the clinical trial or within 31 days of the last study drug dose.
13. Is currently taking a prescription or non-prescription product(s) and food known to be moderate or strong inhibitors or strong inducers (moderate inducers are not prohibited) of cytochrome P450 (CYP3A4), which cannot be discontinued at least 5 half-lives or 14 days prior (whichever is the longer period of time) to Baseline and withheld throughout the clinical study.
14. Has received any experimental or investigational drug, device, or other therapy within 30 days or 5 half-lives (whichever is longer) prior to Screening.
15. Has any of the following abnormal test results at Screening: a serum total bilirubin value >1.5×upper limit of normal (ULN); a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2×ULN. As an exception, participants that present with elevated bilirubin in the absence of elevations in ALT or AST that fits the pattern of Gilbert's syndrome may be enrolled after discussion with the medical monitor and/or sponsor designee if their conjugated bilirubin is below the ULN.
16. History of human immunodeficiency virus (HIV) infection or positive screening result for: HIV 1 or 2 antibodies, hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), or hepatitis C virus antibody (HCVAb).
17. History of long QT syndrome and/or a Fridericia formula corrected QT interval (QTcF) interval >450 msec (males) or >460 msec (females) per electrocardiogram (ECG) done at Screening.
18. Any major psychiatric disorder, including but not limited to depression and anxiety, that is uncontrolled (for the past 90 days) or, in the investigator's judgment, can interfere with any of the study procedures.
19. Has a lifetime history of any suicide attempt, or suicidal ideation with intent within the past 2 years prior to Screening.
20. Participants who have a history of malignancy, myeloproliferative or lymphoproliferative disorders within the past 5 years prior to screen are excluded.

    Exceptions:
    * Participants with completely excised non-melanoma skin cancer (such as basal cell carcinoma or squamous cell carcinoma) or cervical carcinoma in situ are permitted at any time.
    * Participants with a history of other malignancies deemed cured by adequate treatment are also permitted at any time.
21. Has any other significant disease or disorder including but not limited to uncontrolled seizure or epilepsy, diabetes, cardiovascular disease, renal disease, laboratory abnormalities, or environmental factor that, in the opinion of the investigator or sponsor designee, may either put the participant at risk due to participation in the clinical trial, may influence or confound the result of the clinical trial, or may affect the participant's ability to participate in the clinical trial. Uncontrolled epilepsy or seizure is exclusionary and is defined as a seizure or epilepsy diagnosed by a medical clinician and a documented seizure or change in seizure medication (medication or dose) in the last 2 years. An estimated glomerular filtration rate (eGFR) of <60 using the 2021 Chronic Kidney Disease-Epidemiology (CKD-EPI) formula mL/min/1.73m2 or urine albumin creatinine ratio (uACR) of ≥ 30 mg/g is exclusionary.
22. Participant has a positive alcohol or drug screening (including cannabis and cannabis-derived products). The participant can be enrolled in the study, if they are willing to stop use of cannabis or cannabis-related products after the Screening Visit and have a negative cannabidiol (CBD) screen result at Baseline (Day 1). A positive amphetamine, benzodiazepine or opioid drug screening result could be allowed if it is determined that the result is a false positive (for example caused by another medication), or if the result is due to a documented prescribed medication (for example: benzodiazepine or opioid) that in the opinion of the investigator or sponsor designee, is prescribed for a medical condition that aligns with standard of care, is not associated with substance abuse and the investigator's assessment determines that the medical condition and medication dose is stable and expected to remain stable throughout the trial.
23. History of or evidence of psychogenic tremor
24. Prior participation in an ulixacaltamide clinical trial at any time or other clinical trial evaluating a potential drug for ET in the past 6 months (with the exception of participants with documentation that they received placebo treatment only), with the exception of participants that are currently enrolled in and complete the EOT visit in PRAX-944-222 extension period.

Inclusion Criteria for Direct Enrollment into Study 3 LTSS (Following Closure of Enrollment for Study 1 PD and Study 2 RW)

1. Has a clinical diagnosis of ET confirmed during screening and characterized by postural and action tremor.
2. Women of childbearing potential must undertake pregnancy tests, with a documented negative serum pregnancy test at Screening, negative urine pregnancy tests prior to administration of study drug, throughout the intervention periods (as outlined in the SoA) and at the SFU or ED Visit, as appropriate.
3. Is willing and able to use contraception.
4. Has been assessed as an appropriate and suitable candidate by investigator and has a neurological exam and medical record(s) consistent with ET diagnosis, as confirmed by the ERC central reviewer.

Exclusion Criteria for Direct Enrollment into Study 3 LTSS (Following Closure of Enrollment for Study 1 PD and Study 2 RW)

1. Has a known hypersensitivity to any component of the formulation of the ulixacaltamide.
2. Has trauma to the nervous system within 3 months preceding the onset of tremor.
3. Has a history of unilateral tremor or clinical evidence of another medical, neurological, or psychiatric condition that may explain or cause tremor.
4. Has deep brain stimulator (DBS) that in the investigator's discretion is associated with significant stimulation side effects that could impact participant safety.
5. Has a history of substance use disorder consistent with Diagnostic and Statistical Manual of Mental Disorders Fifth Edition Text Revision (DSM-5-TR) criteria. Participants with a previous diagnosis of substance use disorder who have been in remission for at least 2 years can participate in the trial.
6. Is currently pregnant or breastfeeding or is planning to become pregnant during the clinical trial or within 31 days of the last study drug dose.
7. Has received any experimental or investigational drug, device, or other therapy within 30 days or 5 half-lives (whichever is longer) prior to Screening.
8. Has any of the following abnormal test results at Screening: a serum total bilirubin value >1.5×upper limit of normal (ULN); a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2×ULN.
9. History of or active human immunodeficiency virus (HIV) infection or positive screening result for: HIV 1 or 2 antibodies. Evidence of active hepatitis B or hepatitis C infection.
10. History of or currently comorbid long QT syndrome and/or a Fridericia formula corrected QT interval (QTcF).
11. Any major psychiatric disorder, including but not limited to depression and anxiety, that is uncontrolled (for the past 90 days).
12. Has a lifetime history of any suicide attempt, or suicidal ideation with intent within the past 2 years prior to Screening.
13. Participants who have a history of malignancy, myeloproliferative or lymphoproliferative disorders within the past 5 years prior to screen are excluded.
14. Has any other significant disease or disorder including but not limited to uncontrolled seizure or epilepsy, diabetes, cardiovascular disease, renal disease, laboratory abnormalities, or environmental factor.
15. Participant has a positive drug screening associated with drug abuse or misuse.
16. History of or evidence of psychogenic tremor.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Parallel Design: Change from Baseline (CFB) to Week 8 (Day 56) on mADL11 score | 8 weeks (56 days)
  Modified Activities of Daily Living 11 (mADL11) is a composite sum of items 1 to 11 of the TETRAS-ADL subscale. The impact to each function is rated on a 5-point Likert scale from 0 to 4. Before calculating the total score, a scoring adjustment is applied to each item score. The modified score is calculated as the sum of all 11 items (with scoring adjustments) and ranges from 0 to 33 where larger values represent increased direct tremor impact to activities of daily living.
Randomized Withdrawal: The proportion of participants that maintain response, as defined by change in mADL11 score, following randomized withdrawal | 12 weeks (84 days)
  Modified Activities of Daily Living 11 (mADL11) is a composite sum of items 1 to 11 of the TETRAS-ADL subscale. The impact to each function is rated on a 5-point Likert scale from 0 to 4. Before calculating the total score, a scoring adjustment is applied to each item score. The modified score is calculated as the sum of all 11 items (with scoring adjustments) and ranges from 0 to 33 where larger values represent increased direct tremor impact to activities of daily living.
  Change in patient response will compare the proportion of patients in the ulixacaltamide and placebo arm who maintain response based on RW baseline established at Week 8 (Day 56) following randomized withdrawal.
Long-term Safety Study: Number of participants with Adverse Events (AE) and their severity. | Up to 3 years
  The number of participants with Adverse Events (AE) will be reported by preferred term

SECONDARY OUTCOMES:
Parallel Design: Rate of Disease improvement as Measured by mADL11 | 12 weeks (84 days)
  Compare the rate of disease improvement through Day 84 of ulixacaltamide and placebo arms, as measured by the slope of mADL11 over time.
Parallel Design: PGI-C Change at Week 8 (Day 56) | 8 weeks (56 Days)
  PGI-C assesses the participant's change in condition since baseline. The participant is required to assess their condition relative to Baseline (Pre-dose on Day 1) on a 7-point scale from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the participant believes the change is drug-related or not.
Parallel Design: CGI-S Change from Baseline to Week 8 (Day 56) | 8 weeks (56 Days)
  CGI-S assesses the clinician's impression of the participant's current illness state. The clinician should use his/her total clinical experience with this patient population and rate the current severity of the participant's ET on a 7-point scale from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Randomized Withdrawal: Rate of Disease Improvement as Measured by Slope of mADL11 from Day 56 to Day 84 | 4 weeks (28 days)
  Compare the rate of disease improvement from Day 56 to Day 84 of ulixacaltamide and placebo arms.
Randomized Withdrawal: PGI-C at Day 84 | 4 weeks (28 days)
  PGI-C assesses the participant's change in condition. The participant is required to assess their condition relative to Baseline on a 7-point scale from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the participant believes the change is drug-related or not.
Randomized Withdrawal: CGI-S Change from RW Baseline (Day 56) to Day 84 | 4 weeks (28 days)
  CGI-S assesses the clinician's impression of the participant's current illness state. The clinician should use is/her total clinical experience with this patient population and rate the current severity of the participant's ET on a 7-point scale from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).

CONTACTS AND LOCATIONS:
Overall Officials: Director, Clinical Development, Study Director — Praxis Precision Medicines
Locations (1):
- United BioSource LLC, Morgantown, West Virginia, United States